CLINICAL TRIAL: NCT06670079
Title: Prolonged Exposure Therapy to Treat Posttraumatic Stress Disorder in Pregnant Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Kelly Peck, Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVM CHRMS STUDY00002930
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Posttraumatic Stress Disorder; Pregnancy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolonged exposure therapy + incentives for therapy session attendance (Experimental)
  Interventions: Behavioral: Prolonged exposure therapy + incentives for therapy session attendance

INTERVENTIONS:
Behavioral: Prolonged exposure therapy + incentives for therapy session attendance — Prolonged exposure therapy plus incentives for therapy session attendance

SUMMARY:
The goal of this clinical trial is to learn if a treatment for adults with PTSD called prolonged exposure + incentives (PE+) works to treat pregnant patients. The main question it aims to answer is:

Does PE+ decrease PTSD symptoms?

All participants will receive PE+ to see if their PTSD symptoms at the end of the trial are less than at the beginning.

Participants will:

* Receive individual PE+ therapy for 1 hour weekly for 12 weeks.
* Receive financial incentives for attending each PE+ session.
* Attend assessment visits every 4 weeks for the 12 weeks of the trial.
* Allow research staff to collect some information about their labor and delivery from their medical records after their babies are born.

ELIGIBILITY:
Inclusion Criteria:

* Female
* >18 years old
* Gestational age ≤ 25 weeks
* Meet current DSM-5 posttraumatic stress disorder criteria based on the Clinician Administered PTSD Scale for DSM-5
* Participants receiving psychotropic medications must be maintained on a stable dose for >14 days prior to enrollment.

Exclusion Criteria:

* Male
* Under 18 years old
* Gestational age > 25 weeks
* No current diagnosis of PTSD
* Current delusions or hallucinations, unstable bipolar disorder, imminent risk for suicide as assessed by the Mini International Neuropsychiatric Interview
* Enrolled in another ongoing evidence-based treatment for PTSD.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Disorder Symptom Severity - Clinician Rated | From baseline to the 12-week assessment
  Change in posttraumatic stress disorder symptom severity as measured by Clinician Administered PTSD Scale (CAPS-5) for clinician-rated posttraumatic stress symptoms. The CAPS-5 is a 30-item structured interview. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 PTSD symptoms, each with severity scores ranging from 0-4. The overall total severity score for CAPS-5 ranges from 0-80, with lower scores representing better outcomes (less severe PTSD).
Acceptability of prolonged exposure therapy + incentives for therapy session attendance | From baseline to the 12-week assessment
  Change in treatment acceptability as measured by the Treatment Acceptability/Adherence Scale (TAAS). The TAAS is a 10-item scale, each with a range of 1-7 and some of which are reverse-scored. The total TAAS score is calculated by summing the score for the 10 TAAS items and the overall TAAS score ranges from 10-70, with higher scores representing better outcomes (greater treatment acceptability).

SECONDARY OUTCOMES:
Change in posttraumatic stress disorder symptom severity - self-reported | From baseline to the 12-week assessment
  Change in posttraumatic stress disorder symptom severity as measured by PTSD Checklist for DSM-5 (PCL-5) for self-reported posttraumatic stress symptoms. The PCL-5 is a 20-item self-report measure that assesses the 20 symptoms of PTSD. The rating scale is 0-4 for each symptom/item, and overall scores range from 0-80, with lower scores representing better outcomes (less severe PTSD).
Mean change in subjective units of distress | Within 1-hour
  The mean change in subjective units of distress scale (SUDS) ratings from before each imaginal exposure exercise to the peak (highest) level of distress reported during the exercise measured with a single item (range: 0-100).
Mean percent change in heart rate | Within 1-hour
  The mean percent change in heart rate from before each imaginal exposure exercise to peak (highest) heart rate during the exercise
Change in self-reported posttraumatic stress disorder symptom severity between PE sessions | In the 1 week
  The percentage of participants who have a reliable exacerbation in PTSD symptoms between sessions
Prolonged exposure therapy discontinuation | From baseline to the 12-week assessment
  The percentage of participants who complete <8 prolonged exposure therapy sessions
Neonatal birth weight | Delivery
  Neonatal birth weight in grams
Gestational age at delivery | Delivery
  Gestational age at delivery in weeks
Maternal delivery complications | Delivery
  The percentage of participants who experience delivery complications (i.e., abruption/bleeding, hypertensive disorders, and preterm premature rupture of membranes or preterm labor)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided